CLINICAL TRIAL: NCT06827626
Title: Tailored Treatment of Insomnia in Social and Health Care Sector Shift Workers in Occupational Health Care
Acronym: Sote-VURHOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Finnish Work Environment Fund (Other); Terveystalo Oyj (Unknown); Joint Authority HUS (Unknown); The Wellbeing Services County of South Ostrobotnia and TT Botnia Oy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4025601
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Insomnia Chronic; Shift Work Sleep Disorder
Keywords: Shift work; Insomnia; Shift work sleep disorder; CBT-I; Occupational Health Services
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (Experimental): Cognitive-Behavioural Therapy for Insomnia (CBT-I) is tailored for shift workers in social and health care sector. CBT-I is delivered individually (six sessions) by trained nurses. It includes behavioral methods (sleep compression tailored for shift work context), cognitive methods, and shift work related sleep hygiene counselling.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Sleep hygiene counselling (Active Comparator): Sleep hygiene counselling is delivered individually (one session) by trained nurses. It includes sleep hygiene instructions tailored to the context of shift work.
  Interventions: Behavioral: Sleep hygiene counselling

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — Cognitive-Behavioural Therapy for Insomnia (CBT-I) includes behavioral methods, cognitive methods, and sleep hygiene counselling.
  Other Names: CBT-I
  Arms: Cognitive Behavioral Therapy for Insomnia
Behavioral: Sleep hygiene counselling — Sleep hygiene counselling includes common instructions to improve sleep.
  Other Names: Sleep hygiene
  Arms: Sleep hygiene counselling

SUMMARY:
The goal of this clinical trial is to evaluate the usefulness of cognitive behavioural therapy for insomnia (CBT-I) tailored to shift workers in the social and health care sector. The study will also learn about the shift workers' experiences of the acceptability and feasibility of CBT-I and investigate which features of shift work and individual characteristics promote or interfere with the effectiveness of the tailored CBT-I.

The main question the study aims to answer is:

• Does CBT-I tailored to shift workers in the social and health care sector improve perceived insomnia severity, insomnia symptoms, mental health and quality of life?

Researchers will compare CBT-I to a control intervention (short sleep hygiene counselling) to see if CBT-I works to treat insomnia in shift workers.

Participants will:

* Participate in the research intervention (CBT-I tailored to the shift work context; six individual sessions) or the control intervention (sleep hygiene counselling; one individual session)
* Complete the measures (sleep diary, actigraphy and questionnaires) at baseline, after the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment.

DETAILED DESCRIPTION:
Disturbed sleep and insomnia are common among shift workers, and disturbed sleep is considered a key factor in other health risks associated with shift work. However, there are no established treatment practices for treating insomnia in shift workers. This study aims to evaluate the effectiveness of Cognitive-Behavioural Therapy for Insomnia (CBT-I) tailored for social and health care sector shift workers whose work includes night shifts. Furthermore, the study will assess the shift workers' experiences of the acceptability and feasibility of CBT-I from their perspective. The study will also examine which features of shift work and employee characteristics promote or interfere with the effectiveness of the tailored CBT-I.

The study is a randomised controlled trial. Participants will be shift workers in the social and health care sector who work in three or two shifts, including night shifts, and have significant insomnia symptoms. Participants will be recruited through occupational health services (OHS) and social media posts. The FIOH study group will carry out the measurements of the participants. Participants will complete the baseline measures (sleep diary, actigraphy and questionnaires) and then will be randomly assigned to receive the research intervention (CBT-I tailored to the shift work context; six individual sessions) or the control intervention (sleep hygiene counselling; one individual session). The interventions will be delivered by the nurses of the participants´ OHS and the FIOH. Participants will complete the follow-up measures after the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment.

The results of the study can be utilised in OHS to guide and treat shift workers with insomnia as part of supporting their work ability.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* working in social and heath care sector
* 3- or 2-shift work including night shift at least once per month
* full time or nearly full time shift work (75-100 %)
* Insomnia Severity Index score > 10
* duration of insomnia symptoms at least 3 months
* shift work continuing for at least the next year
* sufficient Finnish language skills (coaching materials in Finnish only)

Exclusion Criteria:

* non-assessed or untreated clinically significant somatic or mental symptoms or illnesses or other sleep disorders that could explain current insomnia symptoms
* earlier participation to CBT-I
* other ongoing or planned psychotherapeutic/psychological intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean of Insomnia Severity Index at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Insomnia Severity Index (ISI) contains seven items about insomnia during the last month [item scale 0 (not at all) -4 (very severe)]. The sum of the scores serves as the ISI score.

SECONDARY OUTCOMES:
Change from baseline in means of insomnia symptoms assessed by sleep diary at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Insomnia symptoms are assessed by sleep diary. It is completed using a mobile phone app (Experience Sampling Platform - movisensXS - movisens GmbH). The sleep diary contains questions about the timing of the sleep period, sleep onset latency, wake after sleep onset, number of awakenings after sleep onset, sleep quality, time spent in bed, restedness after sleep, use of sleep-promoting medication, working times, recovery from work, naps and their timing. Total sleep time and sleep efficiency are calculated from the responses. The averages will serve as the outcomes. Participants will keep the sleep diary for 1-2 weeks at each measurement period.
Change from baseline in means of insomnia symptoms assessed by actigraphy at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Insomnia symptoms are also assessed using the Actigraphy Link GT9X. Actigraphy recording is conducted for 1-2 weeks at the same time as the sleep diary. From the actigraphy data, we analyse sleep onset latency, wake after sleep onset, total sleep time, sleep efficiency, naps and their timing. The averages will serve as the outcomes.
Change from baseline in shift work disorder case at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Shift-specific questions on insomnia and sleepiness (SS-Q) -questionnaire measures separately sleepiness and insomnia symptoms in three different shifts (morning, evening and night shifts) and while on holiday over two weeks [item scale 1 (never) - 5 (always)]. Shift work disorder (SWD) cases has to report sleepiness and/or insomnia "never" or "rarely" while on holiday and the never or rarely occurring symptom "often" or "always" in connection to some shift type/types. SWD score [0 (no SWD) or 1(SWD case)] is used as outcome.
Change from baseline in mean insomnia reactivity at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The Ford Insomnia Response to Stress Test (FIRST) contains nine items about insomnia reactivity in potentially stressful situations [item scale 1 (not likely) - 4 (very likely)]. The sum of the scores serves as the FIRST score.
Change from baseline in mean of sleep-related dysfunctional cognitions at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Sleep-related Beliefs and Attitudes about Sleep (DBAS-16) -questionnaire contains 16 items to assesses sleep-related dysfunctional cognitions [item scale 0 (strongly disagree) - 10 (strongly agree)]. The average of the scores serve as the DBAS score.
Change from baseline in mean daytime sleepiness at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The Epworth Sleepiness Scale (ESS) contains eight items to measure the subject's general level of daytime sleepiness in different situations [item scale 0 (would never nod off) - 3 (high chance of nodding off)]. The sum of the scores serves as the ESS score.
Change from baseline in mean depression severity at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The Patient Health Questionnaire (PHQ-9) contains nine items to measure depression severity [item scale 0 (not at all) - 3 (nearly every day)]. The sum of the scores serves as the PHQ-9 score.
Change from baseline in mean anxiety disorder symptoms at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The GAD-7 contains seven items measuring the severity of the symptoms of generalised anxiety disorder [item scale 0 (not at all) - 3 (nearly every day)]. The sum of the scores serves as the GAD-7 score.
Change from baseline in mean burnout symptoms at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The Burnout Assessment Tool (BAT-12) contains 12 items measuring burnout symptoms [item scale 1 (never) - 5 (always)]. The average of the scores serves as the BAT-12 score.
Change from baseline in mean quality of life at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  EuroHIS-8 contains 8 items measuring the quality of life [item scale 1 (worst outcome) - 5 (best outcome)]. The sum of the scores serves as the EUROHIS-8 score.
  Power, M. (2003). Development of a common instrument for quality of life. In A. Nosikov & C. Gudex (edit.), EUROHIS: Developing Common Instruments for Health Surveys (145-159). Amsterdam, Holland: IOS Press.
Change from baseline in mean self-rated work ability at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Work ability measure includes an item measuring self-rated work ability (item scale 0 (not at all) - 10 (very good)].
Change from baseline in mean recovery at the end of treatment (12 weeks after the first session) and at 6 months after the end of treatment. | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  The recovery measure includes an item measuring recovery from work [item scale 1 (badly) - 5 (well)]. In this study, recovery is measured separately in four different shifts (morning, day, evening and night shifts).

OTHER OUTCOMES:
Implementation experiences of the interventions | After the end of treatment (12 weeks after the first session)
  Participants' experiences of the implementation of the interventions are assessed using the Acceptability of Intervention Measure, the Intervention Appropriateness Measure, and the Feasibility of Intervention Measure [each with four items and a scale 1 (completely disagree) - 5 (completely agree)]. The average of each measure serves as a acceptability, appropriateness and feasibility measure of implementation.
Global effectiveness of the treatment | After the end of treatment (12 weeks after the first session)
  Participants rate the global effectiveness of the treatment in improving their overall life situation and well-being using a question from the Consumer Reports survey [item scale 1 (not at all) - 7 (decisive impact)].
Demographic and background information about participants´ work and health | From baseline to the end of treatment (12 weeks after the first session) and to the 6 months after the end of treatment.
  Questions about age, gender, marital status, educational level, shift work related issues (e.g. shift schedules and number of different shifts per month), comorbid conditions, medications and chronotype.
Perceived helpfulness and feasibility per treatment session | After each intervention session
  Participants assess perceived helpfulness and feasibility of each treatment session on a rating scale from 0 (not at all helpful/easy) to 100 (extremely helpful/easy) and answers open-questions about helpfulness and feasibility.

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Joint Authority HUS, Helsinki, Uusimaa
  - Finnish Institute of Occupational Health, Helsinki, Uusimaa
  - Terveystalo Oyj, Helsinki, Uusima
  - The Wellbeing Services County of South Ostrobotnia and TT Botnia Oy, Seinäjoki

IPD SHARING:
Plan to Share IPD: No
Study participants do not give informed consent to have their IPD published (anonymised).

REFERENCES:
- [Result] Ell J, Bruckner HA, Johann AF, Steinmetz L, Guth LJ, Feige B, Jarnefelt H, Vallieres A, Frase L, Domschke K, Riemann D, Lehr D, Spiegelhalder K. Digital cognitive behavioural therapy for insomnia reduces insomnia in nurses suffering from shift work disorder: A randomised-controlled pilot trial. J Sleep Res. 2024 Dec;33(6):e14193. doi: 10.1111/jsr.14193. Epub 2024 Mar 14. PMID 38485134
- [Result] Seligman ME. The effectiveness of psychotherapy. The Consumer Reports study. Am Psychol. 1995 Dec;50(12):965-74. doi: 10.1037//0003-066x.50.12.965. PMID 8561380
- [Result] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Result] Hadzibajramovic E, Schaufeli W, De Witte H. Shortening of the Burnout Assessment Tool (BAT)-from 23 to 12 items using content and Rasch analysis. BMC Public Health. 2022 Mar 22;22(1):560. doi: 10.1186/s12889-022-12946-y. PMID 35313849
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Result] Morin CM, Vallieres A, Ivers H. Dysfunctional beliefs and attitudes about sleep (DBAS): validation of a brief version (DBAS-16). Sleep. 2007 Nov;30(11):1547-54. doi: 10.1093/sleep/30.11.1547. PMID 18041487
- [Result] Kalmbach DA, Pillai V, Arnedt JT, Drake CL. Identifying At-Risk Individuals for Insomnia Using the Ford Insomnia Response to Stress Test. Sleep. 2016 Feb 1;39(2):449-56. doi: 10.5665/sleep.5462. PMID 26446111
- [Result] Vanttola P, Puttonen S, Karhula K, Oksanen T, Harma M. Prevalence of shift work disorder among hospital personnel: A cross-sectional study using objective working hour data. J Sleep Res. 2020 Jun;29(3):e12906. doi: 10.1111/jsr.12906. Epub 2019 Aug 14. PMID 31410909
- [Result] Natale V, Plazzi G, Martoni M. Actigraphy in the assessment of insomnia: a quantitative approach. Sleep. 2009 Jun;32(6):767-71. doi: 10.1093/sleep/32.6.767. PMID 19544753
- [Result] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Result] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- See also: Project web page — https://www.ttl.fi/en/research/projects/tailored-treatment-of-insomnia-in-social-and-health-care-sector-shift-workers-in-occupational-health